CLINICAL TRIAL: NCT01216280
Title: Efficacy and Tolerability Study of Natura-Alpha in the Treatment of Patients With Active Ulcerative Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Natrogen Therapeutics International, Inc (Industry)
Responsible Party: Longgui Wang/President, Natrogen Therapeutics International, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTI-2009-UC1; 70984 (Other: Food and Drug Administration)
Record Dates: First submitted 2010-09-02; First posted 2010-10-07 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-07

CONDITIONS: Ulcerative Colitis
Keywords: Natura-alpha; ulcerative colitis; cytokines; Th1; Th17
MeSH Terms: conditions — Colitis, Ulcerative | interventions — N-methyl-delta-3,3-dihydroindole-2,2 diketone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 x 10 mg placebo capsule (Placebo Comparator): 2 x 10 mg placebo capsules, administered orally with water, b.i.d.
  Interventions: Drug: placebo capsule
- 10mg Natura-alpha + 10 mg placebo (Experimental): 10 mg Natura-alpha capsule + 10 mg placebo capsule administered orally with water, b.i.d.
  Interventions: Drug: 10 mg Natura-alpha capsule and 10 mg placebo capsule
- 2 x 10 mg Natura-alpha capsules (Experimental): 2 x 10mg Natura-alpha capsules administered orally with water, b.i.d.
  Interventions: Drug: 2 x 10 mg Natura-alpha capsules

INTERVENTIONS:
Drug: placebo capsule — 2 x 10 mg placebo capsules administered orally with water, b.i.d.
  Other Names: Group 1
  Arms: 2 x 10 mg placebo capsule
Drug: 10 mg Natura-alpha capsule and 10 mg placebo capsule — 10 mg Natura-alpha capsule and 10 mg placebo capsule administered orally with water, b.i.d.
  Other Names: Group 2
  Arms: 10mg Natura-alpha + 10 mg placebo
Drug: 2 x 10 mg Natura-alpha capsules — 2 x 10mg Natura-alpha capsules administered orally with water, b.i.d.
  Other Names: Group 3
  Arms: 2 x 10 mg Natura-alpha capsules

SUMMARY:
This study is to evaluate the efficacy and tolerability of multiple oral doses of Natura-alpha capsule administered to patients with active ulcerative colitis. This will be a randomized, double-blind, placebo-controlled, parallel-design study. Up to 75 patients will complete this study (20 to 25 patients per treatment group) at approximately 10-12 clinical sites in the Unites States. Patients will be assigned at a 1:1:1 ratio to receive placebo, Natura-alpha 10 mg or Natura-alpha 20 mg, b.i.d. Replacement patients may be added, pending Sponsor approval, if it appears that less than 60 patients will complete the study.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, parallel-design study. Eligible patients will have moderate to severe ulcerative colitis, defined as:

* A Disease Activity Index (DAI) score of 6 to 10 (inclusive);
* Endoscopic evidence of active ulcerative colitis (DAI mucosal appearance sub score of ≥2) as assessed by flexible sigmoidoscopy unless colonoscopy is clinically indicated;
* Rectal bleeding (DAI sub score of ≥1);
* Physician's Global Assessment (PGA) of moderate disease (DAI sub score ≥2). Patients will be randomized to receive placebo, 10 mg Natura-alpha or 20 mg Natura-alpha. Patients will self-administer their assigned dose orally for 28 consecutive days, twice per day (b.i.d) at approximately 8:00 am and 8:00 pm.

The effectiveness and safety of Natura-alpha will be evaluated at baseline, and after 7, 14 and 28 days of treatment. Additional follow-up measurements will take place 7 and 28 days post cessation of treatment (Day 35 and Day 56, respectively). Stool samples for fecal calprotectin (FC) tests and optional blood samples (15 ml) for cytokine tests will be collected and analyzed at sponsor-selected sites and lab for exploratory analyses to be performed at a later date.

Clinical response will be assessed by the Physician's Global Assessment (PGA) on the basis of sigmoidoscopy (Walkiewicz, Werlin et al. 2008) and mucosal appearance (DAI category). Sigmoidoscopy including histopathological examination to assess disease severity and changes in tissue inflammation will be conducted before and after treatment (Day 1, Day 28) by the same endoscopist at each site and read by one sponsor selected central pathologist. Truelove-Richards histological grading system will be applied for disease histological scoring (Pullan, Rhodes et al. 1994; Zhong, Huang et al. 2005; Liang and Ouyang 2008). Safety labs and adverse events (AEs) will be monitored for the duration of the study (including the 7 day follow up visit).

ELIGIBILITY:
Inclusion Criteria:

* Females must be of non-childbearing potential evidenced by being surgically sterile, postmenopausal for at least 12 months or be using acceptable contraception methods.
* Subject is require to meet one of the following criteria:

  1. Newly diagnosed patients with moderate to severe ulcerative colitis evidenced by endoscopy and histopathology, who have never been medically treated for ulcerative colitis, or
  2. Patients with moderate to severe disease, as defined by a Disease Activity Index (DAI) score of 6-10 (inclusive) at the Baseline Visit (assessed at screening and verified at Day 1), with a negative evaluation of the terminal ileum within 3 years of the screening visit, or
  3. Patients with active ulcerative colitis who are refractory or intolerant to therapies of 5-ASA, steroids, immunosuppressants or anti-TNF-alpha.
* Endoscopic evidence of active mucosal disease as assessed by flexible sigmoidoscopy, with a DAI mucosal appearance sub score ≥ 2.
* DAI rectal bleeding sub score of ≥ 1.
* Physician's Global Assessment (PGA) DAI sub score ≥ 2.
* Ability to adhere to the study visit schedule and other protocol requirements.
* Ability to provide voluntary written informed consent.
* Adequate cardiac, renal and hepatic function as determined by site principal investigator and demonstrated by screening laboratory evaluations, and questionnaires, and physical examination results that are within normal limits.

Exclusion Criteria:

* History of colonic or rectal surgery.
* Pregnant or breast-feeding.
* Diagnosis of diabetes, heart failure, unstable angina, hepatic cirrhosis, kidney failure, or any other unstable medical condition.
* Known hypersensitivity to Natura alpha or any of the drug excipients.
* Active and chronic infections.
* Severe ulcerative colitis indicated by Disease Activity Index score > 10.
* Patients with ulcerative proctitis (disease limited to less than 15 cm from the anal verge).
* Use of any vaccine or any other immunostimulator within 4 weeks prior to the screening visit. .
* Use of > 2.4 gm mesalamine or equivalent within 2 weeks prior to the screening visit.
* Use of oral corticosteroids for more than 3 days during the two weeks prior to the screening visit.
* Use of corticosteroid or 5-ASA enemas, foams, or suppositories at any time within two weeks prior to the screening visit. .
* Use of TNF-alpha antibody or any other biologic therapy within 2 months prior to the screening visit. .
* Use of immunosuppressive drugs at any time within four weeks prior to the screening visit. .
* Use of oral or parenteral antibiotics at any time within two weeks prior to the screening visit.
* Diagnosis of Crohn's disease.
* Diagnosis of indeterminate colitis (inability to distinguish between ulcerative colitis and Crohn's disease).
* Diagnosis of microscopic colitis (collagenous or lymphocytic colitis).
* Diagnosis of ischemic, infectious (e.g., salmonella, shigella, etc.), or amebic colitis, or gonococcal proctitis.
* Diagnosis of Clostridium difficile colitis.
* History of positive serology to hepatitis B or C or human immunodeficiency virus (HIV) infection.
* Active alcohol or drug abuse.
* Known malignancy or history of malignancy that would reduce life expectancy.
* Current smoker, or has been a smoker within 6 months prior to the screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Physician's Global Assessment(PGA) | Day 28 after the treatment
  The primary efficacy endpoint will be the proportion of patients in all treatment groups with clinical response (improvement) at Day 28.

SECONDARY OUTCOMES:
Physician's Global Assessment (PGA) | Day 28 after the treatment
  The proportion of patients in all treatment groups who achieve clinical remission at Day 28
Physician's Global Assessment (PGA) | Day 7
  The proportion of patients in all treatment groups who demonstrate clinical response
Physician's Global Assessment (PGA) | 14
  The proportion of patients in all treatment groups who demonstrate clinical response
Physician's Global Assessment (PGA) | Day 28
  The proportion of patients in all treatment groups who demonstrate clinical response who were previously corticosteroid, 5-aminosalicylic acid (5-ASA), immunosuppresant, TNF-alpha antibody therapy-refractory or intolerant
Safety | Day 28
  adverse events, changes in physical examination findings, vital signs, concomitant medications, and laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Longgui Wang, MD, Study Director — Natrogen Therapeutics International, Inc
Locations (10):
- United States (10):
  - Advanced Clinical Research Institute, Anaheim, California
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - AGA Medical Research Associates, LLC, Egg Harbor, New Jersey
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Consultants for Clinical Research, Fairfield, Ohio
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Wisconsin Center for Advanced Research, LLC, Milwaukee, Wisconsin